CLINICAL TRIAL: NCT00361101
Title: Multicenter, Dose-finding Safety and Activity Study of AMD11070 in HIV-infected Patients Carrying X4-tropic Virus.
Brief Title: A Study of AMD11070 in HIV-infected Patients Carrying X4-tropic Virus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD11070-1001
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infections; X4 Tropic Virus
Keywords: HIV; X4 tropic virus
MeSH Terms: conditions — HIV Infections | interventions — mavorixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AMD11070 — 200 mg PO BID (by mouth two times per day) for 10 days.

SUMMARY:
The purpose of this study is to determine the safety and activity of AMD11070 in HIV-infected patients carrying X4-tropic virus.

DETAILED DESCRIPTION:
AMD11070 is a new chemical entity that inhibits HIV-1 entry by binding specifically and reversibly to CXCR4, a coreceptor required by T-tropic virus for membrane fusion and entry into cells. The purpose of this study is to evaluate the safety and relative antiretroviral activity of AMD11070 in HIV-infected individuals who have demonstrated X4 -tropic virus in their plasma. With the ongoing development of other fusion and entry inhibitors and the need for alternative treatment options in patients (especially those with multidrug resistant virus), the demonstration of activity and safety of AMD11070 represents a potentially important advance in antiretroviral therapeutics. This will be the first study that determines the therapeutic potential of anti-CXCR4 compounds in HIV-infected patients.

Note: Study was previously suspended due to non-clinical reports of hepatotoxicity and histologic findings. Study has been completed.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, as documented by any licensed ELISA test kit (confirmed by Western Blot), HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, cDNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
* Both antiretroviral treatment-naïve and -experienced patients. Treatment-experienced patients currently on antiretroviral therapy are required to have a washout period of at least 14 days prior to study entry.
* Presence of X4 tropic virus as determined by a luciferase activity of ≥2000 rlu on the HIV-1 coreceptor tropism assay from a sample collected no more than 56 days prior to study baseline.
* Peripheral blood CD4+ cell count ≤200 cells/mm^3.
* Plasma HIV-1 RNA ≥5000 copies/ml by any standard assay.
* Laboratory values prior to study entry: A. Absolute neutrophil count (ANC) ≥750/mm^3. B. WBC ≥1500/mm^3. C. Hemoglobin ≥10g/dL. D. Platelet count ≥80,000/mm^3. E. Creatinine ≤ 1.2 x ULN. F. AST (SGOT), ALT (SGPT), and alkaline phosphatase ≤ 1.5 x ULN. G. Total bilirubin ≤ 1.2 x ULN. Note: Except for patients who are on atazanavir or indinavir during screening. For these patients, total bilirubin ≤ 4.0 x ULN will be permitted. H. Serum lipase within normal limits. I. PT and PTT ≤ 1.2 x ULN. J. Calcium and magnesium within normal limits.
* Female patients of reproductive potential must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/ml performed within 24 hours before study entry and initiation of the protocol-specified medication..
* All patients must agree not to participate in the conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization).
* Willingness of female patients to discontinue hormonal contraception 1 week prior to study entry. Note: Female patients who discontinue hormonal contraception prior to study entry may resume hormonal contraception after study day 11.
* Karnofsky performance score ≥90 at screening.
* Ability and willingness of patient or legal guardian/representative to give written informed consent.

Exclusion Criteria:

* Patients with a known sensitivity to AMD11070 and its excipients (cellulose, croscarmellose, sodium stearyl fumarate, silicone dioxide, calcium phosphate dihydrate,sodium lauryl sulfate).
* Pregnancy or breast-feeding.
* Any antiretroviral treatment within 14 days prior to study entry.
* Any immunizations within 30 days prior to study entry.
* Treatment with radiation therapy or cytotoxic chemotherapy agents or immuno-modulating agents within 30 days prior to study entry.
* Use of contraindicated prescription medications, herbal supplements, or aspirin within seven days prior to study entry.
* Use of any CYP-3A4 inhibitors or inducers, and P-gp inducers and inhibitors. Use of CYP-450 substrates are allowed in the protocol with the exception of CYP-2D6 and CYP-2C8 substrates.
* Use of any investigational drug (i.e. drugs not approved for any indication) within 30 days prior to study entry.
* Evidence of active infection or acute illness of any kind within 14 days prior to study entry,including HIV-associated opportunistic infection.
* Chronic diarrhea defined as >3 stools/day for more than 4 weeks prior to study entry.
* Documented history of cardiac conduction abnormalities, cardiac arrhythmias, or cardiomyopathy, any repolarization delay (QTc >500msec) or a history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia).
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Any other medical or psychological condition that might, in the opinion of the site investigator, interfere with participation in the study or put the patients at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-10; Primary Completion 2006-08 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
safety and antiviral activity of AMD11070 administered in HIV-infected patients who harbor-X4-tropic virus. | 10 days
the proportion of patients per cohort who have a ≥1 log10 rlu reduction in X4-tropic virus and to describe changes from baseline to Day 10 in log10 rlu corresponding to X4-tropic virus. | 10 days

SECONDARY OUTCOMES:
the relationship between standard pharmacokinetic (PK) measures, viral response, and a shift in T-cell receptor tropism. | 10 days
the relationship of coreceptor tropism phenotype to CD4+ count, viral load, and drug resistance in the screening patient population. | 10 days
the virologic activity of AMD11070 at day 10 of study treatment by analyzing the proportion of patients with Plasma HIV-1 RNA levels <400 and <50 copies/ml and the proportion with a >1 log10 decline in plasma HIV from baseline. | 10 days
changes in CD4+ cell counts and percentages on and off AMD11070. | 10 days
change from baseline in CD34+ cells | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (2):
- Orlando, Florida, United States
- London, United Kingdom

REFERENCES:
- [Result] Moyle G, DeJesus E, Boffito M, Wong RS, Gibney C, Badel K, MacFarland R, Calandra G, Bridger G, Becker S; X4 Antagonist Concept Trial Study Team. Proof of activity with AMD11070, an orally bioavailable inhibitor of CXCR4-tropic HIV type 1. Clin Infect Dis. 2009 Mar 15;48(6):798-805. doi: 10.1086/597097. PMID 19193109